CLINICAL TRIAL: NCT03819556
Title: Swedish Study of Immunotherapy for Milk Allergy in Children
Acronym: SWITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Christina West, Associate professor/Principal investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F07
Record Dates: First submitted 2018-04-20; First posted 2019-01-28 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Milk Allergy
Keywords: Cow milk allergy; Oral immune therapy; Basophil activation test; IgE; Microbiome; Quality of life
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Milk Proteins

STUDY DESIGN:
Intervention Model Description: Open randomized interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active immunotherapy with milk protein (Active Comparator): Daily dose fresh milk protein increased in 11 steps
  Interventions: Other: Milk protein in fresh milk
- Control (No Intervention): Diet free from milk protein

INTERVENTIONS:
Other: Milk protein in fresh milk — Milk protein in increasing doses.
  Arms: Active immunotherapy with milk protein

SUMMARY:
This trial is a two-armed open randomized controlled trial in children aged 5-15 years with challenge proven Immunoglobulin E (IgE)-associated milk allergy.The purpose is to determine if oral immunotherapy with milk can induce tolerance to milk. The active intervention is intake of increasing amounts of fresh milk for six months followed by three years of maintenance treatment with milk. The control group continues their elimination (milk free) diet. The trial will recruit patients at ten pediatric departments in Sweden, coordinated by Umeå University. The primary outcome is milk tolerance (defined as a negative double-blind placebo-controlled milk challenge) at trial completion 3.5 years after start of treatment. Secondary outcomes include allergic symptoms during treatment documented as certain allergic manifestations, changes in immunological and microbial biomarkers, quality of life and nutritional status.

DETAILED DESCRIPTION:
The underlying hypothesis is that exposure to milk in a controlled way can be delivered safely and induce tolerance to milk.The aim of this trial is to evaluate a specific protocol for oral milk intake to achieve sustainable tolerance.

Before randomization all patients are tested for milk allergy using a double-blind placebo-controlled milk challenge and baseline laboratory analyses (specific IgE). Patients with confirmed, challenge-proven milk allergy are randomized to oral immunotherapy (active group) or milk-free diet (control group).The active group will receive a stepwise increase in oral milk intake. The increased dose will be given in hospital outpatient clinics by experienced study staff following a standard protocol. All other doses are given att home where the patients have adrenaline ready to use. When the patient has reached a daily intake of 100 ml of milk without serious allergic reactions they will be maintained on this dosis for three years. At this stage (after finished dose escalation or after six months for the control group) the patients will be tested for the second set of laboratory analyses.

During maintenance, the patients in the active group are encouraged not to avoid milk protein and instead eat milk-containing food when it is offered. Patients in the control group receive standard care with exclusion of milk from their diet for the whole trial duration.

After three years of maintenance therapy for the active group, both groups avoid milk for one week and then undergo a double-blind placebo-controlled milk challenge and the third set of samples for immunological comparison.

The immunological markers are Immunoglobulins (E, G4, A), microbiota and basophilic activation. All patients are also evaluated for quality of life and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Immunoglobulin E (IgE) milk >0.1 kU/L
* Allergic reaction within 2 hours after intake of milk protein
* Age 5-15 years

Exclusion Criteria:

* Uncontrolled asthma, >12 % increase in Forced Expiratory Volume in 1 second (FEV1) after inhaled bronchodilatator and Asthma Control Test (ACT)<20
* No allergic reaction at a controlled milk challenge
* Cancer
* Severe immune deficiency
* Autoimmune disease
* Chronic urticaria
* Eosinophil esophagitis
* Pregnancy and breastfeeding
* Ongoing immunotherapy to one or more allergens

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants that achieve tolerance to milk | 3.5 years after start of treatment
  Tolerance is defined as absence of IgE-mediated allergic symptoms connected to a double-blind placebo-controlled milk challenge

SECONDARY OUTCOMES:
Changes in level of basophil activation (CD sens) in blood | At baseline, after 6 months, after 3.5 years
  Level of basophil activation at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins
Changes in Quality Of Life: FAQLQ-PF | At baseline, after 3.5 years
  Quality Of Life, reported by questionnaire (FAQLQ-PF) after completion of the intervention (3.5 years) compared to pre-trial baseline level. The scale used is Emotional Impact, Food Related anxiety and Dietary Limitations. Each question of the FAQLQ is answered on a 7-point scale. Total FAQLQ scores and domain scores are calculated by dividing the sum of completed items by the number of completed items. Total FaQLQ and domain scores range from 1 "no impairment" to 7 "maximal impairment". Higher values are a worse outcome (low health related quality of life). Subscale is Health related quality of life (HRQoL summary score=(Emotional Impact subscale score + Food Related anxiety subscale score+Dietary Limitations subscale score)/3.
Changes in nutritional status | At baseline, after 3.5 years
  Body Mass Index (BMI) after completion of the intervention (3.5 years) compared to pre-trial baseline levels
Frequency of treatment-demanding adverse effects | 3.5 years
  Number of events with adrenaline injection within 2 hours after a dose of milk (one or two injections) during step-up and maintenance therapy respectively. Number of events with inhalation of bronchodilatator within 2 hours after a dose of milk during step up and maintenance therapy respectively. Number of participants with two or more events with adrenaline injections during step-up and maintenance respectively. Number of participants with two or more events with inhalation of bronchodilatator during step-up and maintenance therapy respectively. Number of participants with no events of adrenaline injections. Number of participants with no events of inhalation with bronchodilatator.
Changes in level of IgE milk in blood | Baseline, 6 months, 3.5 years
  Level of IgE milk including the components IgE casein, IgE lactoglobulin and lactalbumin at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins
Changes in level of IgG4 milk in blood | Baseline, 6 months, 3.5 years
  Level of IgG4 milk at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins
Changes in level of IgA in saliva | Baseline, 6 months, 3.5 years
  Level of IgA at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins
Changes in overall microbial composition in stools | Baseline, 6 months, 3.5 years
  The overall microbial composition at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins will be assessed using amplicon sequencing
Changes in overall microbial composition in saliva | Baseline, 6 months, 3.5 years
  The microbial composition at baseline, after dose escalation and after maintenance therapy and one additional week free from milk proteins will be assessed using amplicon sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Christina E West, MD,PhD, Principal Investigator — Umeå University
Locations (1):
- Solveig Röisgård, Östersund, Jämtland Härjedalen, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Undecided